CLINICAL TRIAL: NCT05959993
Title: The Effect of Human Care Model-Based Nursing Interventions on Psychosocial Adjustment in Patients With Cardioverter Defibrillator
Brief Title: Human Care Model-Based Nursing Interventions on Psychosocial Adjustment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ozgur Demir Gayretli, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ODGayretli
Record Dates: First submitted 2023-05-31; First posted 2023-07-25 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Outpatients; Defibrillators, Implantable
Keywords: Defibrillator; Human Care Model; Psychosocial Adjustment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group participants underwent six interviews at two-week intervals, during which a hybrid and structured nursing intervention was administered.
  Interventions: Behavioral: Human Care Model Based Nursing Interventions
- Control group (No Intervention): Control group participants were not subjected to a structured nursing intervention.

INTERVENTIONS:
Behavioral: Human Care Model Based Nursing Interventions — The interviews scheduled for the intervention group were organized in accordance with the sub-dimensions of the PAIS-SR scale, and the content of each interview was informed by the 10 improvement processes of HCT.
  Arms: Intervention group

SUMMARY:
The aim of the randomized controlled interventional study was to to evaluate the effect of human care model-based nursing interventions on psychosocial adaptation in patients with cardioverter defibrillator. A study was carried out on a sample of 64 patients who had been implanted with a defibrillator. The intervention group participants underwent six interviews at two-week intervals, during which a hybrid and structured nursing intervention was administered.

DETAILED DESCRIPTION:
Aim: The aim of this research was to investigate the impact of nursing interventions that were Watson's Human Care Model- based nursing interventions on the psychosocial adjustment of patients who have undergone implantable cardioverter defibrillator (ICD) implantation.

Design: The present study employs a randomized controlled design with a pretest-posttest control group, conducted over a period spanning from March 2020 to July 2022.

Methods: The research was carried out utilizing an implantable cardioverter on individuals who met the inclusion criteria and provided consent to participate in the study at an adult cardiology outpatient unit located within a university hospital. A study was carried out on a sample of 64 patients who had been implanted with a defibrillator. The intervention group participants underwent six interviews at two-week intervals, during which a hybrid and structured nursing intervention was administered. The data were gathered utilizing an introductory information form and the Psychosocial Adjustment to Illness-Self-Report Scale (PAIS-SR). The statistical methods employed in the data analysis included the chi-square test, t test for independent groups, Mann-Whitney U test, t test for dependent groups, and Wilcoxon signed-rank test.

ELIGIBILITY:
Inclusion Criteria:

* the patient must be of legal age
* the patient must have undergone ICD implantation at least one month prior
* the patient must possess the ability to comprehend and communicate in Turkish
* the patient must not exhibit any hearing or speech impairments
* the patient must not have received a medical diagnosis of a neurological or psychiatric condition that may impact cognitive function, such as Alzheimer's or schizophrenia
* the patient must possess the capability to operate a computer, telephone, and internet

Exclusion Criteria:

* the patient is less than 18 years old
* the patient has hearing and speech problems
* the patient must have received a medical diagnosis of a neurological or psychiatric condition that may impact cognitive function, such as Alzheimer's or schizophrenia
* the patient must not possess the capability to operate a computer, telephone, and internet
* the patient's refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-01-23 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Increasing the patient's psychosocial adjustment with ICD | 10 week later
  Psychosocial Adjustment to Illness Scale -Self Report (PAIS-SR) scale was used. This scale is a multidimensional scale that evaluates psychosocial adjustment to the disease. There are 7 different subscales of the scale that enable the determination of psychosocial adjustment, and the scale consists of a total of 46 items. These subscales are as follows; Orientation to Healthcare, Vocational Environment, Domestic Environment, Sexual Relationships, Extended family Relationships, Social Environment and Psychological distress. The minimum and maximum scores obtained from the scale are between 0-138. The higher the score, the worse the fit. Scores below 35 from the scale indicate good psychosocial adjustment, scores between 35-51 indicate moderately good psychosocial adjustment, and scores above 51 indicate poor adjustment.

CONTACTS AND LOCATIONS:
Overall Officials: Serap Yıldırım, Associate Professor, Study Director — Ege University
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No